CLINICAL TRIAL: NCT01420991
Title: Brain and Abdominal Aneurysm Study (BAAS)
Brief Title: Brain and Abdominal Aneurysm Study
Acronym: BAAS
Status: Completed | Type: Observational
Sponsor: Mayo Clinic (Other)
Responsible Party: Principal Investigator, James F. Meschia, MD, Mayo Clinic
Other Study IDs: 11-003509
Record Dates: First submitted 2011-08-15; First posted 2011-08-22 (Estimated); Last update posted 2025-04-16 (Actual); Status verified 2025-03

CONDITIONS: Aneurysm
MeSH Terms: conditions — Aneurysm

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

SUMMARY:
Aneurysmal subarachnoid hemorrhage (aSAH) is the most deadly kind of stroke. Each year, 40,000 Americans have SAH. Case-fatality approaches 60% and more than half of those who die do so before reaching the hospital. Most commonly, SAH results from rupture of an intracranial aneurysm. Screening high-risk individuals could identify those at greatest risk and decrease the devastating effect of SAH. Aortic Aneurysm also constitutes a major public health problem with high lethality. Current estimates are that ruptured aortic aneurysm kills 13,000 Americans each year. Screening efforts have effectively lowered mortality from aortic aneurysm rupture but a high proportion of those who die did not have a diagnosis of aortic aneurysm prior to rupture.

The relationship between intracranial and aortic aneurysm has long been recognized, but poorly quantified. Recent genome-wide association studies (GWAS) provide a molecular biological evidence for a shared pathophysiology. The chromosome 9p21 locus confers increased risk for both intracranial aneurysms and aortic aneurysms. These GWAS data, along with linkage data for other susceptibility loci, indicate that individuals and families harboring one type of aneurysm may be at especially increased risk of the other.

The rationale for this project is that opportunistic screening for abdominal aortic aneurysms (AAA) may be warranted in patients who present with aneurysmal subarachnoid hemorrhage. This study is meant to see if the yield of screening in this population is too low to justify its routine use. The investigators plan to systematically screen for AAA in all cases of aSAH presenting to MCH for treatment. If no individual out of 81 consecutively screened cases of aSAH has evidence of AAA, then the investigators can have strong confidence that there is a less than 5% chance of finding an AAA in the patient population.

ELIGIBILITY:
1. Men and women age ≥ 18 years.
2. Diagnosis of intracranial aneurysm secured by magnetic resonance angiography (MRA), computed tomographic angiography (CTA), or catheter-based cerebral angiography.
3. Diagnosis of subarachnoid hemorrhage diagnosed by head CT, brain MRI or lumbar puncture.
4. Provides written informed consent.
5. No know diagnosis of aortic aneurysm
6. No history of prior screening for aortic aneurysm
7. No condition like recent abdominal surgical scar that would preclude abdominal ultrasonography
8. No therapy like abdominal hypothermia pads that would preclude abdominal ultrasonography

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: We will enroll 81 patients who present to MCH with aSAH.
Sampling Method: Non-Probability Sample
Enrollment: 271 (Actual)
Dates: Start 2021-10-11 (Actual); Primary Completion 2024-03-02 (Actual); Study Completion 2024-03-02 (Actual)

PRIMARY OUTCOMES:
Prevalence | day 1
  The primary aim is to determine the proportion of patients who are found to have an AAA at the time of enrollment.

SECONDARY OUTCOMES:
Assessment of functional outcomes at 30 days | 30days
  Functional outcomes will be assessed via telephone at one month post hospital discharge

CONTACTS AND LOCATIONS:
Overall Officials: James Meschia, MD, Principal Investigator — Mayo Clinic
Locations (2):
- United States (2):
  - Mayo Clinic in Florida, Jacksonville, Florida
  - Mayo Clinic in Rochester, Rochester, Minnesota

IPD SHARING:
Plan to Share IPD: No